CLINICAL TRIAL: NCT04625244
Title: Can Video Assisted Therapy Replace In-Person Occupational Therapy After Hand Surgery: a Noninferiority Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carilion Clinic (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Peter J Apel, Orthopedic Hand and Upper Extremity Surgeon, Carilion Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-865
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-04

CONDITIONS: Thumb Osteoarthritis
Keywords: video assisted therapy; CMC arthroplasty; carpometacarpal arthroplasty; thumb surgery; hand surgery; home therapy; self directed therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: In-person therapy (No Intervention): Standard of care, in-person therapy with a Certified Hand Therapist (CHT)
- Group 2: Home therapy program (Experimental): Participants will be sent video links to three therapy videos demonstrating postoperative recovery exercises, starting 4 weeks after surgery.
  Interventions: Other: Video assisted home therapy

INTERVENTIONS:
Other: Video assisted home therapy — Subjects will follow along with prerecorded therapy videos.
  Arms: Group 2: Home therapy program

SUMMARY:
This study will investigate a video assisted, home therapy program where participants complete hand therapy on their own following thumb arthroplasty. In this program, participants will receive prerecorded informational videos. Half of the participants in this study will do standard of care, in-person therapy. The other half will be enrolled in the home therapy program. Participants will fill out an assessment of their physical ability before surgery and again three months after surgery. These assessments will be compared between groups. The study team hypothesizes that the video-assisted, home therapy program will be noninferior to traditional in-person therapy.

DETAILED DESCRIPTION:
Current postoperative hand therapy regimens can be burdensome to patients and non-compliance rates are high. Our service area has a lack of hand therapists in the rural areas and the most common barrier to receiving care is access and transportation. In-person therapy requires patients to have significant flexibility in transportation, work schedule and childcare. Travel time and distances put patients who are already disadvantaged at an increased risk of failed treatment. Furthermore, our hand therapy clinics have high utilization after first CMC arthroplasty (thumb joint replacement) procedures, for which therapy is protocol-driven and results are predictable-two aspects that lend this procedure to amenable results from a virtual, unsupervised program.

This study's central hypothesis is that video assisted therapy can be used in postoperative hand therapy without a change in subject outcomes. In this study, the investigators choose to study therapy for one of the most common postoperative diagnoses seen in Carilion Clinic's hand therapy clinics: thumb arthroplasty (replacement of a thumb joint).

Specific Aim 1 is to determine if a video-assisted, home therapy program (pre-recorded instructional videos) can effectively replace in-person occupational therapy for thumb arthroplasty.

Hypothesis: Outcomes of a therapy program consisting of pre-recorded instructional videos will be noninferior to the standard of care regimen for thumb arthroplasty.

The significance of this study is that it investigates a home therapy solution that the investigators expect to increase access to healthcare in rural populations. This study is novel because it will be the first prospective, randomized control trial to investigate the utility of video-assisted home therapy following hand surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective carpometacarpal (CMC) arthroplasty (CPT code 25447)
* Access to a cellphone, tablet or home computer that is connected to internet and has a 5.5" or larger screen

Exclusion Criteria:

* Bilateral procedures
* Revision procedures
* All concomitant procedures, except MCP fusion, CTS release, and thumb trigger finger release
* Artificial CMC joint replacement
* Inability to provide informed consent for the study
* Non-native English speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
Upper extremity function, as assessed by the change in Patient-Reported Outcomes Measurement Information System (PROMIS) v. 2.0 Upper Extremity assessment. | Change from baseline to Day 90 after surgery.
  Improvement in PROMIS upper extremity score from baseline. PROMIS scores are translated into t-scores and range from 0 (worst possible function) to 100 (best possible function). Positive improvement values indicate improvement in function. Negative values indicate a decline in function.

SECONDARY OUTCOMES:
Upper extremity function, as assessed by the change in Patient-Reported Outcomes Measurement Information System (PROMIS) v. 2.0 Upper Extremity assessment. | Change from baseline to Day 365 after surgery.
  Improvement in PROMIS upper extremity score from baseline. PROMIS scores are translated into t-scores and range from 0 (worst possible function) to 100 (best possible function). Positive improvement values indicate improvement in function. Negative values indicate a decline in function.
Pain interference, as assessed by the change in Patient-Reported Outcomes Measurement Information System (PROMIS) v. 1.0 Pain Interference 6a. | Change from baseline to Day 90 after surgery.
  Difference in PROMIS pain interference score from baseline. PROMIS scores are translated into t-scores and range from 0 (minimum pain interference) to 100 (maximum pain interference). Negative differences from baseline indicate improvement in pain interference. Positive differences from baseline indicate worsening of pain interference.
Pain interference, as assessed by the change in Patient-Reported Outcomes Measurement Information System (PROMIS) v. 1.0 Pain Interference 6a. | Change from baseline to Day 365 after surgery.
  Difference in PROMIS pain interference score from baseline. PROMIS scores are translated into t-scores and range from 0 (minimum pain interference) to 100 (maximum pain interference). Negative differences from baseline indicate improvement in pain interference. Positive differences from baseline indicate worsening of pain interference.
Grip strength | Change from baseline to Day 90 after surgery.
  Improvement in grip strength from baseline in operative hand. Measured in pounds force with a dynamometer. A positive change indicates gain of strength.
Key pinch strength | Change from baseline to Day 90 after surgery.
  Improvement in key pinch strength from baseline in operative hand. Measured in pounds force with a dynamometer. A positive change indicates gain of strength.
3-finger pinch strength | Change from baseline to Day 90 after surgery.
  Improvement in 3-finger pinch strength from baseline in operative hand. Measured in pounds force with a dynamometer. A positive change indicates gain of strength.
Thumb radial abduction | Change from baseline to Day 90 after surgery.
  Improvement in thumb radial abduction from baseline in operative thumb. Measured in degrees with a goniometer. A positive change indicates gain of motion.
Thumb palmer abduction | Change from baseline to Day 90 after surgery.
  Improvement in thumb palmer abduction from baseline in operative thumb. Measured in degrees with a goniometer. A positive change indicates gain of motion.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Apel, MD, PhD, Principal Investigator — Carilion Clinic Department of Orthopaedics / Virginia Tech Carilion School of Medicine
Locations (1):
- Carilion Clinic Orthopaedic Surgery, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srikesavan C, Williamson E, Cranston T, Hunter J, Adams J, Lamb SE. An Online Hand Exercise Intervention for Adults With Rheumatoid Arthritis (mySARAH): Design, Development, and Usability Testing. J Med Internet Res. 2018 Jun 27;20(6):e10457. doi: 10.2196/10457. PMID 29950288
- [Background] Hoogland J, Wijnen A, Munsterman T, Gerritsma CL, Dijkstra B, Zijlstra WP, Annegarn J, Ibarra F, Zijlstra W, Stevens M. Feasibility and Patient Experience of a Home-Based Rehabilitation Program Driven by a Tablet App and Mobility Monitoring for Patients After a Total Hip Arthroplasty. JMIR Mhealth Uhealth. 2019 Jan 31;7(1):e10342. doi: 10.2196/10342. PMID 30702438
- [Background] Lee DJ, Calfee RP. The Minimal Clinically Important Difference for PROMIS Physical Function in Patients With Thumb Carpometacarpal Arthritis. Hand (N Y). 2021 Sep;16(5):638-643. doi: 10.1177/1558944719880025. Epub 2019 Oct 18. PMID 31625400